CLINICAL TRIAL: NCT07364760
Title: The Effect of Wellness Coaching and Mobile Application Given To Women Newly Diagnosed With Breast Cancer on Their Psychosocial Adjustment to The Disease and Their Well-Being
Brief Title: The Effect of Group and Mobile Wellness Coaching Given to Women With Breast Cancer on the Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Eylul Yesilyurt, Research Assistant, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Supportive Care
Other Study IDs: SaglikBilimleriU-002
Record Dates: First submitted 2025-09-17; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer Females
Keywords: Breast Cancer; Mobile Application; Wellness Coaching; Psychosocial Adaptation; Wellness
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The study sample will be determined according to inclusion and exclusion criteria. The study groups will consist of 124 individuals who meet the inclusion criteria and have approved the consent form. Patients accepted to participate in the study will be assigned to four groups: Experimental Group 1 Mobile App Wellness Coaching Program group, Experimental Group 2 Group Wellness Coaching Program group, Experimental Group 3 Mobile App + Group Wellness Coaching Program group, and a control group. To avoid bias, participants will be randomly selected according to the order of their arrival.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental Group 1 (Experimental): Patients assigned to Experimental Group 1 will be administered a mobile health application. Patients will be given a pre-test of "Descriptive Information," "Information About the Illness," "Psychosocial Adjustment to the Illness-Self-Report Scale," in a room in the outpatient clinic. The mobile health application will then be introduced and downloaded to their phones. The application will be installed on the phone, and the participant will be asked to create a username and password. User registration to the mobile health application will be conducted in the presence of the researcher. Participants will be provided with a Secret Question/Secret Answer feature to access their account if their username or password is forgotten. During this process, participants will be instructed on how to use the mobile health application. Participants will be encouraged to begin using the mobile health application from the first meeting.
  Interventions: Other: Wellness coaching program with mobile application
- Experimental Group 2 (Experimental): Patients assigned to Experimental Group 2 will be initiated through the Group Wellness Coaching program. A pretest will be administered in a designated room for the patients, which includes "Descriptive Information," "Information About the Illness," "Psychosocial Adjustment to the Illness-Self-Report Scale." The researcher conducting the study will participate in Wellness Coaching training provided by the Zenith Well Health Academy and receive a certificate. Following the training, the content of the Wellness Coaching program will be planned in more detail. The planned Wellness Coaching program will then be implemented for eight weeks, once a week, for a total of eight sessions. Each week, patients will receive training through group sessions. Six groups are planned: five in each group and one group of six. At the end of the eighth week, a survey link will be sent to the patients via Google Forms.
  Interventions: Other: Group Wellness Coaching Program
- Experimental Group 3 (Experimental): Patients assigned to Experimental Group 3 will be initiated using the Mobile App + Group Wellness Coaching Program. A pretest will be administered in a designated room to assess the patients' "Descriptive Information," "Information About the Illness," "Psychosocial Adjustment to the Illness-Self-Report Scale." The planned Group Wellness Coaching program will then be implemented once a week for eight weeks, with a total of eight sessions per week. Patients will also have access to the Mobile App Wellness Coaching program. Wellness Coaching training will be provided both through the mobile app and through group sessions. Group sessions will be held weekly with patients. The plan is to create six groups of five and one group of six. At the end of the eighth week, a survey link will be sent to patients via Google Forms. A post-test will be administered by sending the "Psychosocial Adjustment to Illness-Self-Report Scale.
  Interventions: Other: Mobile app and group wellness coaching program
- Group 4 (No Intervention): Participants in the control group will not receive any intervention. Participants will be given a pre-test of "Descriptive Information," "Information About the Illness," "Psychosocial Adjustment to the Illness-Self-Report Scale" in a room in the outpatient clinic. At the end of eight weeks, a survey link will be sent to patients via Google Forms. The "Psychosocial Adjustment to the Illness-Self-Report Scale" will be sent, followed by a post-test. The Mobile App Wellness Coaching program will be introduced and information will be provided through a brochure. Those who wish will have access to the mobile application. Follow-up tests will be conducted at the end of the first and third months. For control tests, the "Psychosocial Adjustment to Illness-Self-Report Scale" will be filled out by sending a survey link via Google Forms.

INTERVENTIONS:
Other: Wellness coaching program with mobile application — Participants will be provided with wellness coaching training via the mobile application.
  Arms: Experimental Group 1
Other: Group Wellness Coaching Program — Participants will be provided wellness coaching training by the researcher in groups of 5-6.
  Arms: Experimental Group 2
Other: Mobile app and group wellness coaching program — Participants will receive wellness coaching training both via the mobile app and in groups of 5-6 people, provided by the researcher.
  Arms: Experimental Group 3

SUMMARY:
It is believed that this study will serve as a model for a Wellness Coaching program delivered to patients newly diagnosed with breast cancer via a mobile application and contribute to the literature. No other studies have been found in the literature examining the effects of a model-based Wellness Coaching program on the psychosocial adjustment to the disease and well-being of patients newly diagnosed with breast cancer. This demonstrates the originality of this study. In all these respects, it is believed that the study will contribute to the literature and serve as a guide for future studies on the subject.

The purpose of this doctoral dissertation is to determine the effects of Mobile Wellness Coaching and Group Wellness Coaching programs on the psychosocial adjustment to the disease and well-being of women newly diagnosed with breast cancer.

DETAILED DESCRIPTION:
Breast cancer is among the most common types of cancer worldwide. While more common in women, it can also occur in men. According to WHO data, 2.3 million women were diagnosed with breast cancer worldwide in 2022, resulting in 670,000 deaths. The International Agency for Research on Cancer (IARC) predicts that 1 in 20 women worldwide will be diagnosed with breast cancer, with 3.2 million breast cancer cases and 1.1 million breast cancer-related deaths by 2050. In Turkey, breast cancer ranks first among women. According to cancer statistics from the Ministry of Health, 29.3% of women were diagnosed with breast cancer in 2019. According to GLOBOCAN Turkey data, 23.5% (25,249) of women were newly diagnosed with breast cancer in 2022, while 5.7% (7,360) died from breast cancer. Despite increased survival rates thanks to early diagnosis and treatment options, breast cancer poses a multifaceted crisis for women diagnosed with it. The period between a new diagnosis and the first treatment is one of the most stressful times for women with breast cancer. It affects women's physical, psychological, social, and sexual aspects, creating a significant source of stress. Managing stress in women with new breast cancer is crucial for improving the course of the disease, facilitating treatment compliance, ensuring their adaptation to the disease, and improving their overall well-being. Qualitative and descriptive studies conducted with women diagnosed with breast cancer in the literature have identified complex experiences such as pain, anger, anxiety, and life challenges. Having a coach who can help patients going through this complex and challenging process feel they are not alone and who can share positive examples from similar situations with both the client/patient and their family as a companion can foster healthy behavioral changes, increased treatment engagement, and increased belief in recovery and motivation. In a study conducted by Çınar et al., women with breast cancer received mobile app-based education and individual counseling for 12 weeks regarding breast cancer, symptom diaries, and lifestyle recommendations (adequate and balanced nutrition, regular physical activity, stress management, etc.). It was found that the women's quality of life increased and their stress levels decreased. Another study demonstrated that a spiritual nursing care model improved spiritual well-being and the quality of spiritual care in cancer patients. An examination of these practices reveals that healthcare professionals, especially oncology nurses, naturally act as health coaches in this process. A wellness coaching program also evaluates patients holistically, mentally, physically, and spiritually. The goal of the wellness coaching program is to enhance the well-being of breast cancer patients by focusing on their concerns, such as stress, health and illness, life challenges, acceptance of illness, social relationships, physical appearance, and more.

Today, mobile technologies are an important tool for interacting with individuals. Healthcare professionals worldwide have begun to use mobile technology as a tool to reach larger audiences and improve their health. Some studies indicate that mobile apps have the potential to intervene in health behavior changes. Therefore, it is important for nurses to incorporate mobile health apps into the nursing process. There are no mobile apps available in the app markets for Android and iOS operating systems that include a Wellness Coaching program. This thesis aims to provide wellness coaching to patients diagnosed with breast cancer through a mobile app and in person.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older,
* Having recently been diagnosed with breast cancer,
* Not having attended any coaching training since being diagnosed with breast cancer,
* Being fluent in Turkish,
* Literate patients,
* Owning a smartphone.

Exclusion Criteria:

* Being under 18 years of age,
* Refusing to participate in the study,
* Having a visual or hearing impairment,
* Being unable to use a smartphone,

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
pre-test application | 1st month
  First follow-up before intervention A pre-test will be administered to participants before the intervention. Patients who agree to participate in the study will be administered the "Descriptive Information," "Information About the Disease," "Psychosocial Adjustment to the Illness-Self-Report Scale," pre-tests in a room in the outpatient clinic. "Psychosocial Adjustment to Illness-Self-Report Scale" The scale consists of 46 items, including subscales for adjustment to healthcare, occupational environment, family environment, sexual relationships, extended family relationships, social environment, and psychological pressure. The minimum score on the scale is 0, and the maximum is 138. Scores below 35 indicate good psychosocial adjustment, scores between 35 and 51 indicate moderate psychosocial adjustment, and scores above 51 indicate poor psychosocial adjustment. A Wellness Self-Assessment Form will be administered. Participants will be asked to rate the 8 sub-levels of We

SECONDARY OUTCOMES:
final test application | 8th week
  Post-intervention At the end of the eight-week period, a survey link will be sent to patients via Google Forms. A post-test will be administered by sending the "Psychosocial Adjustment to Illness-Self-Report Scale." A Wellness Self-Assessment Form will be administered. Participants will be asked to rate the 8 sub-levels of Wellness (physical, social, emotional, spiritual, etc.) on a scale of 0 to 10. 0 means 'not good at all/bad'. 10 means 'excellent/balanced'. For the follow-up tests, the "Psychosocial Adjustment to Illness-Self-Report Scale" will be sent via Google Forms, and the questionnaire will be completed.Psychosocial Adjustment to Illness-Self-Report Scale: The scale consists of 46 items, including subscales for adjustment to healthcare, occupational environment, family environment, sexual relationships, extended family relationships, social environment, and psychological pressure. The minimum score on the scale is 0, and the maximum is 138. Scores below 3
3rd follow-up | 12th week
  At the end of the first month, patients will be sent a survey link via Google Forms. They will be asked to complete the "Psychosocial Adjustment to Illness - Self-Report Scale" and the "Wellness Self-Assessment Form".
4th follow-up | 20th week
  At the end of the first month, patients will be sent a survey link via Google Forms. They will be asked to complete the "Psychosocial Adjustment to Illness - Self-Report Scale" and the "Wellness Self-Assessment Form".

IPD SHARING:
Plan to Share IPD: Yes
We can share whatever data the journal editor wants to publish.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Result] Ghorbani M, Mohammadi E, Aghabozorgi R, Ramezani M. The effect of applying Spiritual Care Model on well-being and quality of care in cancer patients. Support Care Cancer. 2021 May;29(5):2749-2760. doi: 10.1007/s00520-020-05781-7. Epub 2020 Sep 29. PMID 32995997
- [Result] Lally RM. Acclimating to breast cancer: a process of maintaining self-integrity in the pretreatment period. Cancer Nurs. 2010 Jul-Aug;33(4):268-79. doi: 10.1097/NCC.0b013e3181d8200b. PMID 20467302
- [Result] Mendiola MF, Kalnicki M, Lindenauer S. Valuable features in mobile health apps for patients and consumers: content analysis of apps and user ratings. JMIR Mhealth Uhealth. 2015 May 13;3(2):e40. doi: 10.2196/mhealth.4283. PMID 25972309
- [Result] Sherman DW, Haber J, Hoskins CN, Budin WC, Maislin G, Shukla S, Cartwright-Alcarese F, McSherry CB, Feurbach R, Kowalski MO, Rosedale M, Roth A. The effects of psychoeducation and telephone counseling on the adjustment of women with early-stage breast cancer. Appl Nurs Res. 2012 Feb;25(1):3-16. doi: 10.1016/j.apnr.2009.10.003. Epub 2010 May 6. PMID 20974079
- [Result] Wheaton N, Lenehan J, Amir LH. Evaluation of a Breastfeeding App in Rural Australia: Prospective Cohort Study. J Hum Lact. 2018 Nov;34(4):711-720. doi: 10.1177/0890334418794181. Epub 2018 Sep 20. PMID 30235043
- See also: Related Info — https://www.iarc.who.int/news-events/breast-cancer-cases-and-deaths-are-projected-to-rise-globally/
- See also: Related Info — https://hsgm.saglik.gov.tr/depo/birimler/kanser-db/Dokumanlar/Istatistikler/Turkiye_Kanser_Istatistikleri_2019.pdf
- See also: Related Info — https://gco.iarc.who.int/media/globocan/factsheets/populations/792-turkiye-fact-sheet.pdf.
- See also: Related Info — https://www.who.int/news-room/fact-sheets/detail/breast-cancer

DOCUMENTS (1):
  • Informed Consent Form (2025-09-24): https://cdn.clinicaltrials.gov/large-docs/60/NCT07364760/ICF_000.pdf